CLINICAL TRIAL: NCT07394426
Title: A Phase I, Dose-escalation, Randomized, Single-blind, Placebo-controlled Trial to Evaluate the Safety, Reactogenicity, and Immunogenicity of PepGNP-ChikV, a Synthetic Nanoparticle-based T Cell Next-generational Vaccine Against Chikungunya in Healthy Adults
Brief Title: A Phase I Study of PepGNP-ChikV in Healthy Volunteers
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Gylden Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: GYL-ChikV-101
Record Dates: First submitted 2026-01-26; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Chikungunya; Chikungunya Fever; Chikungunya Virus Infection; Chikungunya Virus Infections; Chikungunya Virus
Keywords: Infectious disease, chikungunya, T cell priming vaccine, first in human, healthy volunteer
MeSH Terms: conditions — Chikungunya Fever; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Dose escalation
Who Masked: Participant
Masking Description: Sponsor will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): PepGNP-ChikV vaccine: 0.28 nmol, 0.83 nmol, 2.5 nmol and 7.5 nmol of total peptide
  Interventions: Biological: PepGNP-ChikV
- Placebo (Placebo Comparator): Placebo (sterile WFI)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PepGNP-ChikV — PepGNP-ChikV vaccine will be administered by an intradermal microneedle device
  Arms: Active
Biological: Placebo — Placebo (sterile WFI) will be administered by an intradermal microneedle device
  Arms: Placebo

SUMMARY:
This is a Phase I, randomized, single-blind, placebo-controlled, study of four separate dose cohorts, with a 42-day interval between each vaccine dose, of a novel Chikungunya Peptide Immunotherapy Vaccine in Healthy Adults (18-60 years of age).

All participants will undergo a screening visit scheduled for a maximum of 28 days before the enrolment in the clinical study and will provide a blood sample for clinical laboratory tests (complete blood count (CBC)*, platelet count, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, serum creatinine and activated partial thromboplastin time (aPTT), human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV)), and a urine sample for tests for Urinary protein, Urinary blood, Urinary glucose and human chorionic gonadotropin β-subunit (βhCG) urine test (only the female participants)) in order to confirm their eligibility for participation in the study.

A total of 40 participants are planned to be enrolled. A randomization system will be used to assign treatment group and participant number at the clinical site.

Participants will receive 2 injections, 42 days apart. A final visit will take place at Day 407 (i.e. 365 days after last vaccination).

Participants will be kept under observation for 30 minutes after each vaccination to ensure their safety. Reactogenicity data will be collected in all participants after each vaccine injection: solicited injection site reactions will be collected for Days 0-10 and Days 42-52 and solicited systemic reactions will be collected for Days 0-21 and Days 42-63. Unsolicited events will be collected for Days 0-52. Serious adverse events (SAEs) will be reported throughout the study (from inclusion until 12 months after last vaccination). Serious and non-serious medically attended adverse events (MAAEs) and adverse events of special interest (AESIs) will be collected throughout the study (from inclusion until 12 months after last vaccination).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals aged ≥18 years to ≤60 years of age, inclusive at time of consent, who are not receiving any excluded concomitant medications as detailed in protocol
2. Informed consent form signed.
3. Determined to be eligible by the Investigator based on medical history, physical examination, and screening laboratory testing.
4. Women of childbearing potential are willing to use effective birth control method(s) for a minimum of 14 days prior to dosing through 90 days after last study vaccination.
5. Male participants with a partner of childbearing potential must agree to use a highly effective method of contraception (e.g. hormonal contraception, intrauterine device, or sterilization) and refrain from sperm donation during the study and for at least 6 months after the last dose of study drug.

Exclusion Criteria:

1. Self-reported or documented history of laboratory-confirmed chikungunya or other mosquito-borne (arthropod) disease, such as Zika or dengue within 90 days prior to consent.
2. Travel in the previous 90 days to areas where exposure to flaviviruses such as Zika, dengue, West Nile Fever are common, as well as areas increasing in cases of chikungunya (refer to the following website: Chikungunya virus disease worldwide overview).
3. Self-reported or documented receipt of any chikungunya (alphavirus) or flavivirus vaccine (investigational or licensed) within 90 days prior to consent.
4. Receipt of any licensed vaccine, including COVID-19 vaccine, within the 28 days prior to consent or planned receipt within 90 days following last study vaccination (if unplanned circumstances subsequent to enrolment necessitate the receipt of a licensed vaccine e.g. tetanus and rabies, in unavoidable clinical settings, these should be documented in the source documents by the Investigator and not considered a protocol deviation. However, if the licensed vaccine is not urgently required, it should be delayed until at least 90 days following last study vaccination).
5. Known systemic hypersensitivity to any of the vaccine components (e.g. gold), or history of a life-threatening reaction to vaccines, or to a vaccine containing any of the same substances.
6. Acute illness according to Investigator judgment especially if febrile (≥38.0°C).
7. Screening laboratory testing reveals a toxicity grading higher than 1 according to Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0 (NCI, 2017). If the Investigator suspects it to be an erroneous result, it can be repeated; the new result should be used for eligibility determination by the Investigator after documenting any clinical significance to any persistently abnormal result.
8. A positive SARS-CoV-2 polymerase chain reaction (PCR) or a positive rapid SARS-CoV-2 antigen test at Screening.
9. Women who are pregnant, or lactating,
10. Calculated body mass index (BMI) > 32.0 kg/m2.
11. Participation in another clinical study investigating a vaccine, drug, medical device, or medical procedure within 90 days or five half-lives, whichever is longer, prior to consent or planned participation in such a study during the period of this clinical study.
12. Receipt of immunoglobulins, blood or blood-derived products within 90 days prior to consent or planned receipt during the period of this chikungunya vaccine study.
13. Known or suspected congenital or acquired immunodeficiency or autoimmune disease; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy, within 90 days prior to consent; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within 90 days prior to consent).
14. Self-reported or documented Hepatitis surface antigen (HBsAg) positivity or antibody against human immunodeficiency virus (HIV), Hepatitis B core, or Hepatitis C. If HIV antibody positive, the participant is to be excluded if HIV is confirmed by further investigation. If Hepatitis C antibody is positive, a Hepatitis C viremia test may be ordered, and, if negative, the participant may continue to be considered for enrolment.
15. Thrombocytopenia (platelet count <150,000/mL) or any coagulation disorder considered clinically significant by the Investigator.
16. Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or study completion.
17. Current alcohol abuse or drug addiction (reported or suspected).
18. Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study or identified as an immediate family member (i.e. parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study. (i.e. in the employment of the clinical study site).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-08-03 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of PepGNP-ChikV candidate vaccine | Onset within 365 days following last vaccination or EOS, whichever is later
  Incidence of serious adverse events (SAEs), medically attended adverse events (MAAEs) and adverse events of special interest (AESIs)
To assess the reactogenicity of PepGNP-ChikV candidate vaccine | Onset within 10 days following each vaccination
  Incidence of solicited local and systemic reactogenicity adverse events (AEs)
To assess the tolerability of PepGNP-ChikV candidate vaccine | Onset within 52 days following each vaccination or End of Study visit (EOS), whichever is later
  Incidence of unsolicited AEs

SECONDARY OUTCOMES:
To determine the CHIKV-specific cellular immune response induced by PepGNP-ChikV | Days 10, 21, 42, 43, 52, 63, 91 and 407 relative to Day 0
  CHIKV-specific immune responses assessed by interferon-gamma (IFN-γ) enzyme-linked immunospot (ELISpot) assays

OTHER OUTCOMES:
To determine the PepGNP-ChikV -specific T cell characterization immune responses | Days 10, 21, 42, 43, 52, 63, 91 and 407 relative to Day 0
  Magnitude, phenotype, and percentage of PepGNP-ChikV peptide (antigen)-specific memory T cells as measured by flow cytometry (including multimers).
To determine the PepGNP-ChikV -specific T cell memory profile immune response | Days 10, 21, 42, 43, 52, 63, 91 and 407 relative to Day 0
  Magnitude, phenotype, and percentage of PepGNP-ChikV peptide (antigen)-specific functional, activation induced T cells as measured by flow cytometry
To check the presence of neutralizing or enhancing antibody responses | Days 1, 10, 21, 42, 43, 52, 63, 91 and 407 relative to Day 0.
  Surrogate Virus Neutralization Tests (sVNTs) to determine neutralizing antibody titres against CHIKV
To check the absence of an antibody mediated response | Days 0 (pre-vaccine), Day 1, Day 10, Day 43 and Day 52
  Magnitude and profiling of expressed, circulating acute cytokine (e.g. IL-1α, Il-1β, IL-1RA, IFN-γ, IFN-α, TNF-α, IL-15 and MCP-1) responses after administration of PepGNP-ChikV vaccine as measured by multiplex platforms (MSD, Luminex)

IPD SHARING:
Plan to Share IPD: No
No plans of IPD currently, as study will be a sponsored clinical study